CLINICAL TRIAL: NCT04017988
Title: A 8 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Ethanol Extracts of Porphyra Tenera(PTE10) on Promotion of Immunity
Brief Title: Efficacy and Safety of Ethanol Extracts of Porphyra Tenera(PTE10) on Promotion of Immunity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JBF-PI-PTE
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Immunity
Keywords: Porphyra Tenera

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethanol Extracts of Porphyra Tenera(PTE10) group (Experimental): 2 times a day, 2 capsules for 1 time, after breakfast/dinner meal (2.512 g/day, Ethanol Extracts of Porphyra Tenera(PTE10) 2.5 g/day)
  Interventions: Dietary Supplement: Ethanol Extracts of Porphyra Tenera(PTE10)
- Placebo group (Placebo Comparator): 2 times a day, 2 capsules for 1 time, after breakfast/dinner meal (2.512 g/day, Ethanol Extracts of Porphyra Tenera(PTE10) 0 g/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ethanol Extracts of Porphyra Tenera(PTE10) — 2 times a day, 2 capsules for 1 time, after breakfast/dinner meal, for 8 week
  Arms: Ethanol Extracts of Porphyra Tenera(PTE10) group
Dietary Supplement: Placebo — Placebo for 8 week
  Arms: Placebo group

SUMMARY:
This study was conducted to investigate the efficacy and safety of ethanol extracts of Porphyra tenera(PTE10) on promotion of immunity

DETAILED DESCRIPTION:
This study was 8 weeks, randomized, double-blind, placebo-controlled human trial. 120 subjects were randomly divided into ethanol extracts of Porphyra tenera(PTE10) group or placebo group. The investigators measure Natural Killer cell activity, Cytokines(IL-2, IL-6, IL-12, IFN-γ, TNF-α), questionnaire scores of upper airway infection.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 50 years over at the screening
* Participants who have fully understood the information provided about the study voluntarily decided to participate and agreed to comply with precautions

Exclusion Criteria:

* Patients whose white blood cell(WBC)<3000/㎕ or >8000/㎕ in the screening examination
* Patients receiving influenza vaccination within 3 months before the screening examination
* Patients who have a body mass index(BMI)<18.5 kg / m^2 or ≥35 kg / m^2 at the screening examination
* Patients with a clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry, musculoskeletal system, inflammatory and hematologic
* Patients who take a medication or health function food that affects your promotion of immunity within 1 month prior to the screening examination
* Patients receiving antipsychotic medication within 3 months prior to the screening examination
* Patients who alcoholic or drug abuse suspected
* Patients who have participated in other clinical trials within 3 months prior to the screening examination
* Patients who show the following relevant results in a Laboratory test

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dl
* Patients who are pregnant or breastfeeding
* Patients who may become pregnant and have not used appropriate contraceptives
* Patients who the principal investigator judged inappropriate for the participant in this study because of a laboratory test result, etc

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes of Natural Killer cell activity | 0 week, 8 week
  Natural Killer cell activity was measured in study baseline and 8 week. A ratio of effector cell and target cell was 50:1, 25:1, 12.5:1.
  (Experimental - Effector Spontaneous - Target Spontaneous) / (Target Maximum - Target Spontaneous) × 100

SECONDARY OUTCOMES:
Changes of Cytokines | 0 week, 8 week
  For blood Cytokines analysis, collect 3 ml of blood in one SST tube for 5 ml, leave at room temperature for 30 minutes for clotting, after then centrifuge at 3000 rpm (or 2000 xg) for 10 minutes.
  Inspection item were IL-2, IL-6, IL-12, IFN-γ, TNF-α.
Changes of Upper respiratory infection questionnaire score | 0 week, 4 week, 8 week
  The upper respiratory infection questionnaire will investigate the occurrence of symptoms of upper respiratory infections (or symptoms), the score by symptom, the duration (days), and survey on the day of visit (1st, 2nd and 3rd visits).
  The questionnaire items were classified into three groups according to whether or not the symptoms of upper respiratory infections (or symptoms) occurrence (yes or no), the types of symptoms (sore throat, rhinorrhea, nasal obstruction, sneezing, hoarseness, myalgia, earache, fever, headache, cough, sputum, dyspnea, diarrhea, nausea, vomiting)and symptoms level (0 if no symptoms, 1 if slightly, 2 if normal, 3 severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea